CLINICAL TRIAL: NCT05639842
Title: Pain in Competitive Athletes With Physical Disabilities: Techniques for Its Management, Support Received and Perceived Difficulties
Brief Title: Pain in Competitive Athletes With Physical Disabilities: Techniques, Support and Perceived Difficulties
Status: Completed | Type: Observational
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Sandra Constantino Murillo, Principal Investigator, Universidad Politecnica de Madrid
Other Study IDs: UPMadrid.
Record Dates: First submitted 2022-11-21; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Pain; Athletes; Physical Disability
Keywords: Athlete; Physical disability; Chronic pain; Psychological models
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pain in competitive athletes with physical disabilities. Techniques for its management, support received and perceived difficulties. — A total of 413 athletes with physical disabilities participated in the study, 157 Spanish athletes and 260 Latin American athletes. The athletes were contacted through different sports federations, Paralympic Committees and sports teams of people with disabilities.For the distribution of the questionnaire, the researcher made an initial telephone contact with the Spanish Paralympic Committee and the Spanish Sports Federation for People with Physical Disabilities, to explain the objectives of the study and ask for their collaboration in the dissemination. Subsequently, the information was officially sent to them by email.

SUMMARY:
Pain in physically disabled athletes affects the sporting career directly or indirectly through psychological consequences. Numerous studies address psychological skills in able-bodied athletes and in able-bodied athletes they are scarce.This information is part of a research project aimed at finding resources to help athletes in their pain management.

DETAILED DESCRIPTION:
The purpose of this study is to determine how competitive athletes perceive how pain can affect their sporting careers; what techniques and/or strategies athletes use for pain management and how useful these are; to determine the extent to which athletes with disabilities have received support for pain management and to what extent they have found it useful; and to determine the difficulties they often face in managing their pain.The aim of this questionnaire is to find out how pain, resulting from injury, can affect the sporting careers of competitive athletes with physical disabilities and what techniques they use to manage it.

ELIGIBILITY:
Inclusion Criteria:

Athletes:

* Competitive athletes.
* Physical disability.
* Age without criteria.

Exclusion Criteria:

* Failure to meet the inclusion criteria.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 413 participants were interviewed on a voluntary basis. Spanish and Latin American nationality.
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-04-17 (Actual)

PRIMARY OUTCOMES:
Cross-sectional surveys | 5 months
  An ad-hoc questionnaire was developed with questions that sought to respond to the specific objectives of this study, taking into consideration the information obtained in the previous qualitative study. The questionnaire consisted of 74 questions, 68 closed multiple-choice and 6 open-ended, organised into six sections: characteristics of the athlete, how pain affects their sporting career, tolerance and acceptance of pain, techniques and strategies for managing pain, social support for pain management and finally difficulties in pain management. A Likert scale from 1 (very infrequently) to 5 (very often) was used.Depending on the interpretation of the questions asked in each section, higher scores mean a better or worse result.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Constantino Murillo, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Sandra Constantino Murillo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No